CLINICAL TRIAL: NCT04897841
Title: Obstetric Liposomal Bupivacaine Via Surgical Transversus Abdominis Plane Block for Post Cesarean Pain Control: a Single-blind Pilot Randomized Controlled Trial
Brief Title: Obstetric Liposomal Bupivacaine Via Surgical Transversus Abdominis Plane Block for Post Cesarean Pain Control
Acronym: OBLiBupi
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Meriter Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UPH-Meriter IRB 2021-005; A532860 (Other: UW Madison); SMPH/OBSTET & GYNECOL (Other: UW Madison); Protocol Version 6/13/2022 (Other: Meriter IRB); 2021-0410 (Other: UW-Madison IRB)
Record Dates: First submitted 2021-05-18; First posted 2021-05-24 (Actual); Results first posted 2023-10-30 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2023-10

CONDITIONS: Cesarean Section Complications; Pain; Opioid Use
Keywords: cesarean
MeSH Terms: conditions — Pain | interventions — Bupivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- control arm (Placebo Comparator): The control arm will receive 30 mL of bupivacaine HCl plus 50 mL of saline injected into the lateral transversus abdominis plane via surgical approach (abdominal approach).
  Interventions: Drug: Bupivacaine Hydrochloride; Other: saline
- Intervention: liposomal bupivacaine (Experimental): The intervention arm will receive 30 mL of bupivacaine HCl plus 30 mL of saline plus 20 mL of liposomal bupivacaine injected into the lateral transversus abdominis plane via surgical approach (abdominal approach).
  Interventions: Drug: Liposomal bupivacaine; Drug: Bupivacaine Hydrochloride; Other: saline

INTERVENTIONS:
Drug: Liposomal bupivacaine — 20 mL prior to closing fascia, the active drug (bupivacaine) is encapsulated in a liposomal platform and released slowly over the course of days with an approximate 72 hour duration.
  Arms: Intervention: liposomal bupivacaine
Drug: Bupivacaine Hydrochloride — 30 mL bupivacaine hydrochloride 0.25 percent, local post-surgical anesthetic
Other: saline — post-surgical saline

SUMMARY:
This study seeks to identify whether the addition of liposomal bupivacaine to regular bupivacaine and saline administered via surgical transversus abdominis plane (TAP) block will reduce the cumulative opioid dose in the first 48 hours after cesarean. 60 women scheduled for cesarean at Unity-Point Health Meriter Hospital in Madison, Wisconsin will be enrolled and can be expect to be on study for up to 6 weeks post-partum.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether liposomal bupivacaine administered via surgical TAP block at the time of Cesarean delivery will reduce the total dose of opioids received. The hypothesis is that liposomal bupivacaine will reduce the total dose of opioids received in the immediate 48 hours post-delivery.

Secondary outcomes will include participant self-reported pain scores, participant-reported incidence of side effects, and development of objective complications such as dysrhythmias. Other outcomes collected will include length of stay, time to first rescue analgesic medication, total dose of opioids at 12, 24, 36, 72 hours and during the hospital stay, use of supplemental oxygen during hospitalization, breastfeeding rates, both exclusive and in combination with formula use, amount of opioid prescribed at discharge and whether refills were requested or administered, rates of chronic pain at six weeks postpartum, and six week Edinburgh Depression Screen scores. Neonatal outcomes such as fetal weight, five-minute Apgar scores and development of adverse outcomes such as neonatal intensive care unit (NICU) admission will also be collected because NICU admission can impact maternal opioid use.

Primary Objective:

* To determine whether liposomal bupivacaine administered via surgical TAP block at the time of cesarean delivery will reduce the total dose of opioids received in the first 48 hours after surgery.
* Hypothesis: The hypothesis is that liposomal bupivacaine administered via surgical TAP block at the time of cesarean delivery will reduce the total dose of opioids received in the first 48 hours after surgery.
* Developmental Sub Aim: If liposomal bupivacaine administered via surgical TAP block does reduce the total dose of opioids received, to determine the degree of the reduction in order to allow for an adequately powered randomized-controlled trial.

Secondary Objective:

* To determine whether liposomal bupivacaine administered via surgical TAP block at the time of cesarean delivery will reduce patient-reported pain scores and opioid-related side effects, including respiratory compromise.
* Hypothesis: The hypothesis is that liposomal bupivacaine administered via surgical TAP block at the time of cesarean will reduce patient-reported pain scores and opioid related side effects.

ELIGIBILITY:
Inclusion Criteria:

* Maternal age greater than or equal to 18
* Singleton or multifetal pregnancy
* Able to receive neuraxial analgesia
* Planned/ scheduled Cesarean delivery OR non-urgent Cesarean delivery at UnityPoint-Health Meriter with adequate time to consider and consent to the study
* Able to provide consent in English

Exclusion Criteria:

* Known hypersensitivity to bupivacaine (defined as a history of a reaction or allergy to bupivacaine (injectable, intravenous, or transdermal) reported by patient or documented in the medical record
* Contraindication to regional analgesia
* Positive urine drug screen at admission to the hospital, if ordered for clinical purposes.
* Current opioid use or opioid use disorder per patient report or documented in the medical record
* Chronic opioid use or opioid use disorder, either patient reported or documented in the medical record, defined as opioid use on most days for greater than 3 months
* Planned cesarean hysterectomy (excluded due to anticipated blood loss and alternative pain control measures, possible prolonged intubation)
* Planned vertical midline incision (excluded due to possible different postpartum pain)
* Presence of renal dysfunction precluding the use of NSAIDs (NSAIDs are part of the usual postpartum pain regimen/ hospital protocol) per discretion of the treating physician or PI
* Ischemic heart disease, congestive heart failure, or cardiomyopathy of pregnancy precluding the use of NSAIDs (NSAIDs are part of the usual postpartum pain regimen/ hospital protocol) per discretion of the treating physician or PI
* Significant liver dysfunction precluding the use of acetaminophen (acetaminophen is part of the usual postpartum pain regimen/ hospital protocol) per discretion of the treating physician or PI
* Coagulopathy
* Planned discharge from the hospital less than 48 hours postpartum
* Unable to receive post-operative scheduled acetaminophen for any reason, such as allergy to acetaminophen or elevated liver function tests precluding acetaminophen use
* Unable to receive post-operative scheduled NSAIDs for any reason, such as allergy to ketorolac or ibuprofen, or renal dysfunction precluding NSAID use
* Seizure disorder: Specifically, poorly controlled seizure disorder defined as having had a seizure within the last three years despite antiepileptic use or poorly managed seizure disorder due to medication non-compliance.
* Cardiac disease or arrhythmia: Defined as ischemic heart disease, peripartum cardiomyopathy, heart failure (with reduced or preserved ejection fraction, compensated or decompensated). Patients with a remote history of non-cyanotic pediatric cardiac surgery (like a VSD closure or PDA ligation as a child) do not need to be excluded. History of adult cardiac surgery without ongoing problems or treatments other than chronic anticoagulation (mitral valve repair for MVP or aortic valve replacement for bicuspid aortic valve for example) would not need to be excluded. History of repaired congenital cyanotic heart disease should be considered for exclusion, ultimately up to the anesthesiologist that day. A patient with a history of arrhythmias not requiring medication or ablation would NOT need to be excluded and could be included in the study. History of ablation or active anti-arrhythmic medication should be considered for exclusion.
* Hypoxia: Defined as requiring supplemental oxygen during the day.
* Acidosis. This will be uncommon in our population, but if someone has active diabetic ketoacidosis will exclude.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-10-11 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-10-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen M Antony, MD, MSCI, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- Unity-Point Health Meriter, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Antony KM, McDonald RC, Gaston L, Hetzel S, Li Z. Surgical transversus abdominis plane block with liposomal bupivacaine at cesarean: a pilot randomized trial. Am J Obstet Gynecol MFM. 2024 Feb;6(2):101273. doi: 10.1016/j.ajogmf.2023.101273. Epub 2023 Dec 26. PMID 38154599

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Arm | Intervention: Liposomal Bupivacaine
Started | 29 | 31
Completed | 29 | 31
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Arm | Intervention: Liposomal Bupivacaine | Total
Number analyzed (Participants) | 29 | 31 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.7 (5.3) | 33.0 (3.8) | 33 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 31 | 60
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 29 | 29 | 58
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 25 | 28 | 53
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 29 | 31 | 60

OUTCOME MEASURES:

1. Primary Outcome: Total Opioid Usage in Oral Morphine Equivalents
Description: Compared via Student's t-test or Mann-Whitney U test if the distribution is non-normally distributed
Time Frame: up to 48 hours postpartum
Measure: Median (Inter-Quartile Range); unit: morphine milligram equivalents
Arm/Group | Control Arm | Intervention: Liposomal Bupivacaine
Number analyzed (Participants) | 29 | 31
morphine milligram equivalents | 8 [0 to 40] | 2 [0 to 24]

2. Secondary Outcome: Median Post-operative Pain Scores Measured on NRS
Description: Numeric rating scale (NRS) which rates pain on a 0-10 scale where 10 is increased pain.
Time Frame: Collected per standard of care every 4-6 hours up to 24 hours postpartum
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Control Arm | Intervention: Liposomal Bupivacaine
Number analyzed (Participants) | 29 | 31
score on a scale | 3.75 [2 to 5] | 3 [2 to 4]

3. Secondary Outcome: Maximum Post-operative Pain Scores Measured on NRS
Description: Numeric rating scale (NRS) which rates pain on a 0-10 scale where 10 is increased pain.
Time Frame: Collected per standard of care every 4-6 hours up to 24 hours postpartum
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Control Arm | Intervention: Liposomal Bupivacaine
Number analyzed (Participants) | 29 | 31
score on a scale
  First 12 hours postpartum | 2.5 [2 to 5] | 2 [1 to 3.5]
  12-24 hours postpartum | 3.5 [2 to 4.5] | 3 [2 to 4.5]

4. Secondary Outcome: Minimum Post-operative Pain Scores Measured on NRS
Description: Numeric rating scale (NRS) which rates pain on a 0-10 scale where 10 is increased pain.
Time Frame: Collected per standard of care every 4-6 hours up to 24 hours postpartum
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Control Arm | Intervention: Liposomal Bupivacaine
Number analyzed (Participants) | 29 | 31
score on a scale
  First 12 hours postpartum | 2 [1.5 to 3.5] | 2 [1 to 2]
  12-24 hours postpartum | 3 [2 to 4] | 3 [2 to 3]

5. Secondary Outcome: Incidence of Opioid Side Effects
Description: Number of patients reporting opioid-related side effects, such as pruritis, constipation, nausea, and mental clouding.
Time Frame: up to 7 days postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Control Arm | Intervention: Liposomal Bupivacaine
Number analyzed (Participants) | 29 | 31
Participants
  Respiratory events | 0 | 0
  Pruritis | 0 | 1
  Constipation | 0 | 0
  Nausea and/or vomiting | 2 | 2
  Mental clouding | 1 | 1

6. Secondary Outcome: Percentage of Participants With Adverse Events
Description: Percentage of complications of bupivacaine, such as local burning, nausea, dizziness, drowsiness, serious skin reactions such as blistering, confusion, blurred vision, ringing in the ears, arrhythmias, methemoglobinemia, and allergies and hypersensitivities
Time Frame: up to 7 days postpartum
Measure: Number; unit: % of participants with adverse events
Arm/Group | Control Arm | Intervention: Liposomal Bupivacaine
Number analyzed (Participants) | 29 | 31
% of participants with adverse events | 10 | 6

7. Secondary Outcome: Time to First Rescue Analgesic Medication
Description: Time to first rescue analgesic medication, measured in minutes from arrival in the post-anesthesia care unit (PACU) until the first as needed opioid dose is administered.
Time Frame: up to 7 days postpartum
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Control Arm | Intervention: Liposomal Bupivacaine
Number analyzed (Participants) | 29 | 31
minutes | 21.8 [5.1 to 29.2] | 18.2 [3.2 to 29.5]

8. Secondary Outcome: Total Dose of Opioids in Oral Morphine Equivalents
Time Frame: at 12, 24, 72 hours postpartum and entire hospital stay
Measure: Median (Inter-Quartile Range); unit: morphine milligram equivalents
Arm/Group | Control Arm | Intervention: Liposomal Bupivacaine
Number analyzed (Participants) | 29 | 31
morphine milligram equivalents
  12 hours postpartum | 0 [0 to 0] | 0 [0 to 6]
  24 hours postpartum | 0 [0 to 8] | 0 [0 to 8]
  72 hours postpartum | 24 [0 to 40] | 6 [0 to 32]
  entire hospital stay | 24 [0 to 40] | 6 [0 to 46]

9. Other Pre Specified Outcome: Length of Postpartum Hospital Stay
Time Frame: up to 7 days postpartum
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Control Arm | Intervention: Liposomal Bupivacaine
Number analyzed (Participants) | 29 | 31
Days | 2.97 [2.76 to 3.81] | 2.82 [2.09 to 3.13]

10. Other Pre Specified Outcome: Incidence of Supplemental Oxygen Use During Hospitalization
Description: Number of participants requiring supplemental oxygen use
Time Frame: up to 7 days postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Control Arm | Intervention: Liposomal Bupivacaine
Number analyzed (Participants) | 29 | 31
Participants | 0 | 0

11. Other Pre Specified Outcome: Number of Participants Breastfeeding at Hospital Discharge
Description: Breastfeeding rates, both exclusive and breastfeeding with supplementation at the time of discharge
Time Frame: up to 7 days postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Control Arm | Intervention: Liposomal Bupivacaine
Number analyzed (Participants) | 29 | 31
Participants
  Exclusive breastfeeding | 26 | 29
  Breastfeeding with supplementation | 3 | 2

12. Other Pre Specified Outcome: Amount of Opioid Prescribed at Discharge
Time Frame: up to 7 days postpartum
Measure: Median (Inter-Quartile Range); unit: number of opioid tablets
Arm/Group | Control Arm | Intervention: Liposomal Bupivacaine
Number analyzed (Participants) | 29 | 31
number of opioid tablets | 10 [0 to 15] | 0 [0 to 10]

13. Other Pre Specified Outcome: Percentage of Participants With Opioid Refills Requested
Time Frame: 6 weeks postpartum
Measure: Number; unit: percentage of participants with refill
Arm/Group | Control Arm | Intervention: Liposomal Bupivacaine
Number analyzed (Participants) | 29 | 31
percentage of participants with refill | 8.33 | 3.6

14. Other Pre Specified Outcome: Number of Opioid Pills Used
Time Frame: 6 weeks postpartum
Measure: Median (Inter-Quartile Range); unit: number of pills used
Arm/Group | Control Arm | Intervention: Liposomal Bupivacaine
Number analyzed (Participants) | 29 | 31
number of pills used | 0 [0 to 3] | 0 [0 to 1.5]

15. Other Pre Specified Outcome: Postnatal Depression Screen
Description: Participants self-reported feeling down or depressed
Time Frame: 6 weeks postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Control Arm | Intervention: Liposomal Bupivacaine
Number analyzed (Participants) | 29 | 31
Participants | 10 | 12

16. Other Pre Specified Outcome: Percentage of Participants Who Would Recommend Treatment
Description: 2 weeks postpartum, participants will be asked to report whether they would recommend the treatment they received
Time Frame: 2 weeks postpartum
Measure: Number; unit: percent who would recommend treatment
Arm/Group | Control Arm | Intervention: Liposomal Bupivacaine
Number analyzed (Participants) | 29 | 31
percent who would recommend treatment | 81.0 | 78.6

17. Other Pre Specified Outcome: 6 Week Postpartum Satisfaction Survey Response Percentage
Description: 6 weeks postpartum, participants will be asked whether they would recommend the treatment they received.
Time Frame: 6 weeks postpartum
Measure: Number; unit: percent who would recommend treatment
Arm/Group | Control Arm | Intervention: Liposomal Bupivacaine
Number analyzed (Participants) | 29 | 31
percent who would recommend treatment | 70.8 | 78.6

18. Other Pre Specified Outcome: Fetal Weight
Time Frame: at birth
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Control Arm | Intervention: Liposomal Bupivacaine
Number analyzed (Participants) | 29 | 31
grams | 3312 (540) | 3395 (448)

19. Other Pre Specified Outcome: Five-minute Apgar Scores
Description: The Apgar Score is a measure of fetal health status immediately after birth. It comprises five components: 1) color, 2) heart rate, 3) reflexes, 4) muscle tone, and 5) respiration, each of which is given a score of 0, 1, or 2 for a total possible score of 0-10, where higher scores indicate better health.
Time Frame: 5 minutes after birth
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Arm | Intervention: Liposomal Bupivacaine
Number analyzed (Participants) | 29 | 31
score on a scale | 8.79 (0.49) | 8.74 (.68)

20. Other Pre Specified Outcome: Number of Participants With at Least One Newborn Admitted to the Neonatal Intensive Care Unit (NICU)
Description: NICU admission is a potential confounding variable for maternal opioid use.
Time Frame: up to 7 days postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Control Arm | Intervention: Liposomal Bupivacaine
Number analyzed (Participants) | 29 | 31
Participants | 5 | 5

21. Other Pre Specified Outcome: Number of Participants Readmitted to the Hospital
Time Frame: up to 6 weeks postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Control Arm | Intervention: Liposomal Bupivacaine
Number analyzed (Participants) | 29 | 31
Participants | 0 | 2

ADVERSE EVENTS:
Time Frame: 6 weeks post-partum
Arm/Group | Control Arm | Intervention: Liposomal Bupivacaine
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/31
Serious Adverse Events (participants affected / at risk) | 1/29 | 1/31
Other Adverse Events (participants affected / at risk) | 8/29 | 7/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Arm (N=29) | Intervention: Liposomal Bupivacaine (N=31)
Post-partum hemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Nystagmus (Eye disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Arm (N=29) | Intervention: Liposomal Bupivacaine (N=31)
Local burning or blistering (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3)
Dizziness (General disorders) | 1 (1) | 2 (2)
Edema, erythema, pruritis, or irritation at site of injection (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Arrythmias (Cardiac disorders) | 1 (1) | 1 (1)
Confusion or tremors (Nervous system disorders) | 1 (1) | 0 (0)
Any potential or definitive local anesthetic systemic toxicity or symptoms (LAST) (Investigations) | 2 (2) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Nausea and vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2)
Mental clouding (General disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-11): https://cdn.clinicaltrials.gov/large-docs/41/NCT04897841/Prot_SAP_000.pdf